CLINICAL TRIAL: NCT04563936
Title: A Multicenter, Randomized, Open-Label Phase Ⅲ Trial to Compare Efficacy and Safety of Goserelin Acetate Sustained-Release Microspheres for Injection (LY01005) and ZOLADEX® in Patients With Prostate Cancer
Brief Title: Efficacy and Safety of LY01005 in Patients With Prostate Cancer Compared to ZOLADEX®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY01005/CT-CHN-302
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; LY01005; Efficacy; Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01005 3.6 mg (Experimental): Intramuscular injections of LY01005 3.6 mg every 28 days for a maximum of 3 consecutive doses.
  Interventions: Drug: LY01005 3.6 mg
- ZOLADEX® 3.6 mg (Active Comparator): Subcutaneous injections of ZOLADEX® 3.6 mg every 28 days for a maximum of 3 consecutive doses.
  Interventions: Drug: ZOLADEX® 3.6 mg

INTERVENTIONS:
Drug: LY01005 3.6 mg — LY01005 was administered as 3 intramuscular (IM) injections, 28 days apart. As concomitant medications, Casodex® (50 mg/day) was orally administered during the whole study period.
  Other Names: Goserelin Acetate Sustained-Release Microspheres for Injection
  Arms: LY01005 3.6 mg
Drug: ZOLADEX® 3.6 mg — ZOLADEX® was administered as 3 Subcutaneous (SC) injections, 28 days apart. As concomitant medications, Casodex® (50 mg/day) was orally administered during the whole study period.
  Other Names: goserelin acetate implant 3.6 mg
  Arms: ZOLADEX® 3.6 mg

SUMMARY:
This is a multicenter, randomized, open-label, active comparator-controlled phase Ⅲ trial to compare efficacy and safety of Goserelin Acetate Sustained-Release Microspheres for Injection (LY01005) and ZOLADEX® in patients with prostate cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active comparator-controlled phase Ⅲ trial using non-inferior design. A total of 290 patients with prostate cancer who were suitable for endocrine therapy were enrolled into the screening period from D-21 to D-10 before administration. Eligible subjects were treated with bicalutamide tablets (Casodex®, 50 mg/day) from D-10 (± 3d) before administration and randomized in a 1:1 ratio to receive LY01005 3.6 mg or ZOLADEX® 3.6 mg after completion of pretreatment. All subjects were administered once every 28 days for three doses until intolerable toxicity, disease progression requiring other anti-tumor treatments, withdrawal of consent, loss to follow-up, death or the end of the whole study. Blood samples were collected at the specified time points of the screening period, before/behind each dose to detect serum testosterone, LH, FSH and PSA. Safety evaluation (including vital signs, physical examination, laboratory tests, 12 ECG, adverse events, etc.) was conducted as required in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years or older.
2. Patients with pathological confirmed prostate cancer suitable for endocrine therapy (except for neoadjuvant endocrine therapy), including those who are suitable for endocrine therapy (such as patients with biochemical recurrence after adjuvant endocrine therapy and radical therapy) following radical therapy.
3. Serum testosterone level ≥ 1.50 ng/mL (5.21 nmol/L) at the screening visit (based on the test results of research centers).
4. Life expectancy of at least 9 months.
5. ECOG score of ≤ 2.
6. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 10^9/L, white blood cell count ≥ 3 x 10^9/L, and hemoglobin ≥ 90 g/L at the screening visit.
7. Total bilirubin (TBIL) ≤ 1.5×ULN, both ALT and AST ≤ 2.5×ULN (or ≤ 5.0×ULN for patients with liver metastases) at the screening visit.
8. Calculated creatinine clearance (Cockcroft-Gault formula) of ≥ 30 mL/min at the screening visit.
9. Patients who voluntarily sign an IRB-approved informed consent form before the screening visit, are willing to abide by the restrictions of the study, and complete the prescribed examinations.

Exclusion Criteria:

1. Patients with prostate cancer who receive previous or ongoing endocrine therapy (surgical castration or other endocrine therapy including GnRH receptor agonists, GnRH receptor antagonists, anti-androgens, estrogens, megestrol acetate, etc.), except for patients with prostate cancer undergoing prostatectomy, radiotherapy or cryotherapy who have received neoadjuvant/adjuvant endocrine therapy for no more than 6 months and discontinued the above therapy more than 6 months before screening.
2. Has received prostatic surgery within 4 weeks prior to the Screening Visit, or plan to receive surgical treatment during the trial.
3. Patients with confirmed or suspected hormone-resistant prostate cancer.
4. Has previously received hypophysectomy or adrenalectomy, or who have pituitary lesions.
5. Has received 5-α reductase inhibitors (finasteride, dutasteride, eridasteride, etc.) within 1 month before the first dose.
6. Has previously received goserelin.
7. Has received an investigational drug, an investigational biological product or an investigational medical device, and discontinued within 1 month or 5 half-lives of the corresponding drug before the screening visit, whichever is longer.
8. History of severe asthma, anaphylaxis, or severe urticaria and/or angioedema.
9. History or presence of another malignancy, other than surgically removed squamous/basal cell carcinoma of the skin, within the last 5 years.
10. History of the following medical histories within 6 months: myocardial infarction, unstable angina, coronary revascularization, New York Heart Association (NYHA) class ≥ II cardiac insufficiency, severe unstable arrhythmia; Or the presence of arrhythmia requiring treatment at the screening period.
11. Hypertensive patients with poor blood pressure control after medication (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg at the screening visit).
12. Has received coumarin anticoagulants.
13. Patients with type 1 diabetes or type 2 diabetes with poor glycemic control (glycosylated hemoglobin > 8% at the screening visit).
14. Has congenital long QT syndrome or QT/QTc interval prolongation (QTc ≥ 450 ms) at the screening visit; Or has received drugs that may prolong QT/QTc interval at the screening visit.
15. Alcoholics, drug addicts or drug abusers.
16. Patients of childbearing potential who refuse using effective contraception during the entire trial.
17. Patients with viral hepatitis B who are taking anti-hepatitis B virus (HBV) drugs or need drug treatment (those who need drug treatment must meet the following 2 conditions at the same time: 1. HBV DNA level: HBeAg-positive patients, HBV DNA ≥ 20,000 IU/ml [equivalent to 10^5 copies/mL]; HBeAg-negative patients, HBV DNA ≥ 2,000 IU/ml [equivalent to 10^4 copies/mL]; 2. ALT ≥ 2 x ULN).
18. Patients who are seropositive for hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) antibody.
19. Known to be allergic to the active ingredients or any excipients of the investigational drug, or other GnRH analogues.
20. Other conditions considered unsuitable for enrollment by the investigator (such as spinal cord compression due to prostate cancer metastatic lesions of pyramid, pulmonary interstitial disease or other serious diseases).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with serum testosterone ≤50 ng/dL (1.735 nmol/L) on Day 29 after the first dose. | Day 29 after the first dose
The cumulative percentage of subjects with the maintenance of serum testosterone ≤50 ng/dL (1.735 nmol/L) from Day 29 to Day 85. | from Day 29 to Day 85

SECONDARY OUTCOMES:
Significant Castration Rate | from Day 29 to Day 85
  The percentage of subjects with serum testosterone ≤20 ng/dL (0.7 nmol/L) on Day 29 after the first dose, and the cumulative percentage of subjects with the maintenance of serum testosterone ≤20 ng/dL (0.7 nmol/L) from Day 29 to Day 85.
The percentage of subjects with an acute increase in serum testosterone above castrate levels within 72 hours following repeated dosing. | within 72 hours following the second and third administration
Percentage changes compared to baseline in serum LH level after administration. | from baseline to Day 85
Changes in serum LH level after administration. | from baseline to Day 85
Percentage changes compared to baseline in serum FSH level after administration. | from baseline to Day 85
Changes in serum FSH level after administration. | from baseline to Day 85
Percentage changes compared to baseline in serum PSA level after administration. | from baseline to Day 85
Changes in serum PSA level after administration. | from baseline to Day 85
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | up to Day 85
Incidence of serious adverse events (SAE). | up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gu C, Wang Z, Lin T, Liu Z, Han W, Zhang X, Liang C, Liu H, Yu Y, Xu Z, Liu S, Wang J, Jia L, Yao X, Liao W, Fu C, Tan Z, He G, Zhu G, Fan R, Yang W, Chen X, Liu Z, Zhong L, Shi B, Ding D, Chen S, Wei J, Yao X, Chen M, Lu Z, Xie Q, Hu Z, Wang Y, Guo H, Fan T, Liang Z, Chen P, Wang W, Xu T, Li C, Xing J, Liao H, He D, Wu Z, Yu J, Feng Z, Yang M, Dou Q, Zeng Q, Li Y, Gou X, Zhou G, Wang X, Zhu R, Zhang Z, Zhang B, Tan W, Qu X, Sun H, Gan T, Ye D. Efficacy and safety of LY01005 versus goserelin implant in Chinese patients with prostate cancer: A multicenter, randomized, open-label, phase III, non-inferiority trial. Chin Med J (Engl). 2023 May 20;136(10):1207-1215. doi: 10.1097/CM9.0000000000002638. Epub 2023 Apr 3. PMID 37010251